CLINICAL TRIAL: NCT03435536
Title: Influence of Pancreatic Adenocarcinoma Excision Surgery on Peripheral and Portal Circulating Tumor DNA: Prospective Exploratory Pilot Study.
Brief Title: Surgery Impact on Circulating Tumor DNA in Pancreatic Cancer
Acronym: ICAPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/17/0327
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2023-01

CONDITIONS: Resectable Pancreatic Cancer
Keywords: circulating tumor DNA; kinetic; pancreatic cancer; pancreatoduodenectomy; Next Generation Sequencing
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Circulating tumor DNA (Experimental): circulating tumor DNA rate at various times of pancreatic cancer resection
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples will be taken to analyze the circulating tumor DNA rate by NGS

SUMMARY:
Pancreatic cancer represents the fourth cause of death by cancer in western countries. The only curative treatment is surgery but this one is possible only in 10 to 15 % of cases. To date, there are few biomarkers in circulating blood as prognostic or diagnostic markers in pancreatic cancer. The purpose of this study is to determine if the pancreatic tumor mobilization during its resection impacts the quantity of circulating tumor DNA in peripheral and portal blood.

DETAILED DESCRIPTION:
The investigators will analyze if the tumor mobilization increases circulating DNA rate in peripheral and portal blood. Moreover, circulating tumor DNA will be measured during 12 months after surgery in peripheral blood. They will use a gene mutation detection technique called Next Generation Sequencing (NGS) which is more specific than a simple Polymerase Chain Reaction (PCR).

ELIGIBILITY:
Inclusion Criteria:

* Every patient taken care by Toulouse University Hospital for the resection of a non-metastatic pancreatic adenocarcinoma by whipple resection.
* Patient aged over 18 years old
* Patient having given his written consent
* Patient with social insurance coverage

Exclusion Criteria:

* Patients who had surgery, but their pathological examination of the resected specimen does not contain adenocarcinoma.
* Patient for whom the surgery was not realized (exploratory laparotomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Kinetic of circulating tumor DNA evaluation in resected pancreatic cancer. | Kinetic up to one year
  To analyse circulating tumor DNA rate in the portal vein and in peripheral blood at various times of pancreatic cancer resection. Kinetic to 1 day before surgery, during surgery and after surgery (1 day, 10days , one month, 3 months, 6 months and one year after surgery)

SECONDARY OUTCOMES:
Overall survival | Kinetic up to one year
  to analyse correlation between circulating tumor DNA rate and overall survival and survival without recurrence. Kinetic to 1 day before surgery, during surgery and after surgery (1 day, one month, 3 months, 6 months and one year after surgery)
Correlation between circulating tumor DNA rate and Ca19.9 dosage | Kinetic up to one year
  to analyse correlation between circulating tumor DNA and Ca19.9 rate after dosage of C19.9. Kinetic to 1 day before surgery, and after surgery (on day, one month, 3 months, 6 months and one year after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel CUELLAR, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maulat C, Canivet C, Cabarrou B, Pradines A, Selves J, Casanova A, Doussine A, Hanoun N, Cuellar E, Boulard P, Carrere N, Buscail L, Bournet B, Muscari F, Cordelier P. Prognostic impact of circulating tumor DNA detection in portal and peripheral blood in resected pancreatic ductal adenocarcinoma patients. Sci Rep. 2024 Nov 8;14(1):27296. doi: 10.1038/s41598-024-76903-y. PMID 39516243